CLINICAL TRIAL: NCT06470360
Title: Clinical Outcomes of Absorbable or Hem-o-lok Clip Closure of the Cystic Stump in Laparoscopic Cholecystectomy: a Prospective Randomised Clinical Trial
Brief Title: Comparison of the Safety of Absorbable and Hem-o-lok Clips in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulas Aday (Other Government)
Responsible Party: Sponsor-Investigator, Ulas Aday, Ass. Prof., Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Organization: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dicle University
Record Dates: First submitted 2024-04-14; First posted 2024-06-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: laparoscopic cholecystectomy; cystic duct closure; safety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single absorbable (Active Comparator): Cystic duct to be closed with absorbable single clip
  Interventions: Other: Surgycal procedure
- Single Hem-o-lok (Active Comparator): Cystic duct to be closed with Hem-o-lok single clip
  Interventions: Other: Surgycal procedure

INTERVENTIONS:
Other: Surgycal procedure — surgical technique

SUMMARY:
Safe closure of the cystic duct is the critical step in laparoscopic cholecystectomy. In the literature, the investigators did not observe any prospective study analysing the use of absorbable single clip and Hem-o-lok single clip. In this prospective study, the reliability of the two methods will be compared using a single clip.

DETAILED DESCRIPTION:
In this prospective randomised controlled clinical study; closure of the cystic duct in laparoscopic cholecystectomy will be performed by two different methods. Early clinical results and long-term effects on neighbouring anatomical structures will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy ASA I-III Patients who accepted the study

Exclusion Criteria:

* open surgery emergency cholecystectomy refuse to trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Complications of patients using absorbable and haem-olok clips will be compared according to the Clavien-Dindo scoring system. | first 30 day
  Is it safe to close the cystic stump with a single (haem-o-lok or absorbable) clip?

SECONDARY OUTCOMES:
The costs of the clips used | one week
  The costs of the clips used will be determined in dollars using Student's t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Duman, Principal Investigator — Kartal Kosuyolu
Locations (1):
- Kartal Koşuyolu Higher Specialization Training and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No